CLINICAL TRIAL: NCT00494897
Title: PETHEMA LAL-RI/96: Treatment for Patients With Standard Risk Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Pethema, pethema
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL-RI/96
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Mercaptopurine; Prednisone; Vincristine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Asparaginase
Drug: Cyclophosphamide
Drug: Cytarabine
Drug: Daunorubicin
Drug: Mercaptopurine
Drug: Prednisone
Drug: Vincristine
Drug: Methotrexate
Procedure: Intrathecally treatment

SUMMARY:
The objective of current protocol is try improve the results of chemotherapy treatment in patients with ALL wich is not indicated the peripheral stem cell transplant in first remission, with an intensive consolidation follow by re-inductions.

DETAILED DESCRIPTION:
Induction therapy:

Patients with standard risk receive vincristine (1,5 mg/m2)IV on days 1, 8, 15 and 22;daunorubicin (30 mg/m2)IV on days 1, 8, 15 and 22; oral or IV prednisone 60 mg/m2/day, days 1 to 27 and 30 mg/m2/day, days 28 to 35;asparaginase 10.000 UI/m2 IM or IV, days 10 to 12, 17 to 19 and 24 to 26;cyclophosphamide (500 mg/m2)IV days 1, 2 and 29; methotrexate, cytosine arabinoside and hydrocortisone, days 1 to 22.

Patients older than 55 years are not treated with asparaginase and cyclophosphamide.

Consolidation therapy (1):

Standard risk: Mercaptopurine 50 mg/m2, PO, days 1 to 7, 28-35 and 56-63; methotrexate (3g/m2)IV/24 hours, day 1, 28 and 56; VM-26 (150 mg/m2)/12 hours, IV, days 14 and 42; ARA-C (500 mg/m2)/12 hours, IV days 14-15 and 42-43; intrathecally treatment, days 1, 28 and 56.

Patients over 50 years: Mercaptopurine (50 mg/m2), PO, days 1 to 7, 28-35 and 56-63;methotrexate (1,5 g/m2) IV/24 hours, day 1, 28 and 56; VM-26 (150 mg/m2)/12 hours, IV days 14 and 42; ARA-C (500 mg/m2)/12 hours, IV days 14-15 and 42-43; intrathecally treatment, days 1, 28 and 56.

Consolidation therapy (2)/Reinduction: one cycle similar to induction. It starts one week after last dose of mercaptopurine.Dexamethasone 10 mg/m2/day,PO or IV, days 1-14 and 5 mg/m2/day, PO or IV days 15-21; VCR: 1,5 mg/m2 IV, days 1, 8 and 15; Daunorubicin 30 mg/m2 IV, days 1, 2, 8 and 9; cyclophosphamide 600 mg/m2/day IV, days 1 and 15; Asparaginase: 10.000 UI/m2 IM or IV, days 1-3 and 15-17;intrathecally treatment days 1 and 15

Maintenance therapy 1:administration of continuous chemotherapy (mercaptopurine and methotrexate) and reinductions until one year from diagnosis.

* Continuous chemotherapy:

  * MP 50 mg/m2/day PO
  * MTX 20 mg/m2/week IM
* Reinductions

  * VCR: 1,5 mg/m2 IV, day 1.
  * PDN: 60 mg/m2/day, IV or PO days 1 to 7
  * L-ASA: 20.000 UI/m2, IM or IV day 1.
  * Intrathecally day 1

Seven cycles, weeks 25, 29, 33, 37, 41, 45 and 49.

Maintenance therapy 2:administration of continuous chemotherapy (mercaptopurine and methotrexate) while second year from diagnosis (weeks 53 to 104).

* MP 50 mg/m2/day, PO
* MTX 20 mg/m2/week, IM.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 15 years) with ALL standard risk no prior antiblastic chemotherapy

Exclusion Criteria:

* Mature B-ALL (FABL3) or with cytogenetic ALL "Burkitt-like" alterations (t[8;14], t[2;8], t[8;22])
* Mixed forms of ALL
* Acute Leukemia no differentiate
* Patients with coronary disorders, valvular or hypertensive cardiopathy
* Patients with chronic liver disorders
* Chronic pulmonary disorders
* Renal insufficiency
* Neurologic disfunctions
* ECOG 3 and 4
* No signed consent form

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 1996-06; Primary Completion 2007-05 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment in adults with standard risk acute lymphoblastic leukemia | 2 years

SECONDARY OUTCOMES:
Demonstrate that in this group of patients, the CNS relapse is not frequently and is not necessary cranial radiotherapy | 2 years
To evaluate the treatment tolerance | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ribera Josep Mª, Dr, Study Director — Germans Trias i Pujol Hospital
Locations (87):
- Spain (87):
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital Ntra. Sra. Sonsoles, Ávila, Avila
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clínic, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital vall d'Hebrón, Barcelona, Barcelona
  - Hospital Valle Hebrón-Materno Infantil, Barcelona, Barcelona
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital Mútua de Terrassa, Terrassa, Barcelona
  - Hospital general de Castellón, Castelló, Castellón
  - Hospital Puerta del Mar, Cadiz, Cádiz
  - Complejo Hospitalario Reina Sofía, Córdoba, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital Juan Ramón Jiménez, Huelva, Huelva
  - Hospital Médico Quirúrgico Ciudad de Jaén, Jaén, Jaen
  - Hospital Juan Canalejo, A Coruña, La Coruña
  - Hospital Arnau de Vilanova, Lleida, Lleida
  - Clínica Puerta de Hierro, Madrid, Madrid
  - Hospital Clínico San Carlos de Madrid, Madrid, Madrid
  - Hospital de Fuenlabrada, Madrid, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid, Madrid
  - Hospital Universitario de la Princesa, Madrid, Madrid
  - Hospital Universitario Princcipe de Asturias, Madrid, Madrid
  - . Hospital Clínico Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital del Río Carrión, Palencia, Palencia
  - Hospital Son Dureta, Palma de Mallorca, Palma de Mallorca
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Joan XXIII, Tarragona, Tarragona
  - Hospital Verge de la Cinta, Tortosa, Tarragona
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital Clínic, Valencia, Valencia
  - Hospital General Universitario, Valencia, Valencia
  - Hospital La Fe, Valencia, Valencia
  - Hospital Meixoeiro, Vigo, Vigo
  - Hospital Clínico Lozano Blesa, Zaragoza, Zaragoza
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital Regional Universitario Infanta Cristina, Badajoz
  - Basurtuko Ospitalea, Basurto
  - Complejo Hospitalario de Cáceres, Cáceres
  - Hospital Nuestra Señora de Alarcos, Ciudad Real
  - Hospital Virgen de la Luz, Cuenca
  - Hospital General de Elda, Elda
  - Institut Català d'Oncologia,, Girona
  - Hospital de San Jorge, Huesca
  - Hospital de Jerez de la Frontera, Jerez de la Frontera
  - Hospital General de Lanzarote, Lanzarote
  - Complejo Hospitalario León, León
  - Complexo Hospitalario Xeral-Calde, Lugo
  - Hospital 12 de Octubre, Madrid
  - Hospital de la Princesa, Madrid
  - Hospital Doce de Octubre, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Althaia, Xarxa Asistencial de Manresa, Manresa
  - H. Carlos Haya, Málaga
  - Hospital General Morales Meseguer, Murcia
  - Hospital Santa María del Rosell, Murcia
  - Hospital Virgen del Castillo de Yecla, Murcia
  - Complejo Asistencial Son Dureta, Palma de Mallorca
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Verge del Toro, Palma de Mallorca
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital Virgen del Camino, Pamplona
  - Complejo Hospitalario de Pontevedra_Hospital Montecelo, Pontevedra
  - Hospital de Sagunto, Sagunto
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital San Pedro de Alcántara, San Pedro
  - Clínica Sant Camil, Sant Pere de Ribes
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital de Santiago de Compostela, Santiago de Compostela
  - Hospital General de Segovia, Segovia
  - H.U. Virgen del Rocio, Seville
  - Hospital Nuestra Señora del Prado, Toledo
  - Hospital Virgen de la Salud, Toledo
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Dr. Peset, Valencia
  - Hospital Francesc de Borja, Valencia
  - Hospital General Básico de la Defensa, Valencia
  - Hospital Clínico de Valladolid, Valladolid
  - Complejo Hospitalario Universitario de Vigo, Vigo
  - Hospital Txagorritxu, Vitoria-Gasteiz
  - Hospital de Galdakao, Vizcaya

REFERENCES:
- [Background] P Bastida, JJ Ortega, ME González-Valentín, C Calvo, J Marín, JM Ribera, M Fontanillas. Tratamiento de la leucemia aguda linfoblástica en niños. Resultados del protocolo PETHEMA 89. Sangre 1996; 41 (supl 3): 94
- [Background] JM Ribera, M Fontanillas, A Oriol, E Feliu, J Maldonado, J Hernández-Rivas, J Marín, J Zuazu, C Rivas, J Alcalá, S Brunet, FJ Rafecas, J Carnero, J Besalduch, S Gardella, J Alvarez, J garcía Conde, F Fernández-Calvo, J Martínez, MJ Moro, R casanova, J Maciá, F Ortega, R Salinas, J varela, JF san Miguel, JJ Ortega. Leucemia aguda linfoblástica (LAL) del adulto. Resultados del protocolo PETHEMA LAL-89. Sangre 1996; 41 (supl 3): 94.
- [Background] Sanz MA, Martin G, Rayon C, Esteve J, Gonzalez M, Diaz-Mediavilla J, Bolufer P, Barragan E, Terol MJ, Gonzalez JD, Colomer D, Chillon C, Rivas C, Gomez T, Ribera JM, Bornstein R, Roman J, Calasanz MJ, Arias J, Alvarez C, Ramos F, Deben G. A modified AIDA protocol with anthracycline-based consolidation results in high antileukemic efficacy and reduced toxicity in newly diagnosed PML/RARalpha-positive acute promyelocytic leukemia. PETHEMA group. Blood. 1999 Nov 1;94(9):3015-21. PMID 10556184
- [Background] Kantarjian HM, Walters RS, Keating MJ, Smith TL, O'Brien S, Estey EH, Huh YO, Spinolo J, Dicke K, Barlogie B, et al. Results of the vincristine, doxorubicin, and dexamethasone regimen in adults with standard- and high-risk acute lymphocytic leukemia. J Clin Oncol. 1990 Jun;8(6):994-1004. doi: 10.1200/JCO.1990.8.6.994. PMID 2189958
- [Background] GIMEMA ALL 0183: a multicentric study on adult acute lymphoblastic leukaemia in Italy. GIMEMA Cooperative Group. Br J Haematol. 1989 Mar;71(3):377-86. PMID 2649141
- [Background] Clarkson B, Gaynor J, Little C, Berman E, Kempin S, Andreeff M, Gulati S, Cunningham I, Gee T. Importance of long-term follow-up in evaluating treatment regimens for adults with acute lymphoblastic leukemia. Haematol Blood Transfus. 1990;33:397-408. doi: 10.1007/978-3-642-74643-7_75. PMID 2182430
- [Background] Lluesma-Gonalons M, Pavlovsky S, Santarelli MT, Eppinger-Helf M, Dorticos Bavea E, Corrado C, Carnot J. Improved results of an intensified therapy in adult acute lymphocytic leukemia. Ann Oncol. 1991 Jan;2(1):33-9. doi: 10.1093/oxfordjournals.annonc.a057821. PMID 2009234
- [Background] Tomonaga M, Omine M, Morishima Y, Hirano M, Dogi H, Imai K, et al. . Individualized induction therapy followed by intensive consolidation and maintenance including asparaginase in adult ALL: JALSG-ALL87 study. Haematologica 1991; 76 (suppl 4): 68
- [Background] Smedyr B, Simonsson B, Björkholm M, Carneskog J, Gahrton G, Grimfors G, et al. Treatment of adult acute lymphoblastic and undifferentiated (ALL/AUL) leukemia according to a national protocol in Sweden. Haematologica 1991; 76 (suppl 4): 107.
- [Background] Ellison RR, Mick R, Cuttner J, Schiffer CA, Silver RT, Henderson ES, Woliver T, Royston I, Davey FR, Glicksman AS, et al. The effects of postinduction intensification treatment with cytarabine and daunorubicin in adult acute lymphocytic leukemia: a prospective randomized clinical trial by Cancer and Leukemia Group B. J Clin Oncol. 1991 Nov;9(11):2002-15. doi: 10.1200/JCO.1991.9.11.2002. PMID 1941059
- [Background] Cuttner J, Mick R, Budman DR, Mayer RJ, Lee EJ, Henderson ES, Weiss RB, Paciucci PA, Sobol R, Davey F, et al. Phase III trial of brief intensive treatment of adult acute lymphocytic leukemia comparing daunorubicin and mitoxantrone: a CALGB Study. Leukemia. 1991 May;5(5):425-31. PMID 2033963
- [Background] Stryckmans P, De Witte T, Marie JP, Fillet G, Peetermans M, Bury J, Muus P, Andrien JM, Hayat M, Jaksic B, et al. Therapy of adult ALL: overview of 2 successive EORTC studies: (ALL-2 & ALL-3). The EORTC Leukemia Cooperative Study Group. Leukemia. 1992;6 Suppl 2:199-203. No abstract available. PMID 1578934
- [Background] Bassan R, Battista R, Rohatiner AZ, Love S, Carter M, Buelli M, Viero P, D'Emilio A, MacCallum P, Amess J, et al. Treatment of adult acute lymphoblastic leukaemia (ALL) over a 16 year period. Leukemia. 1992;6 Suppl 2:186-90. PMID 1578929
- [Background] Hoelzer D, Thiel E, Ludwig WD, Loffler H, Buchner T, Freund M, Heil G, Hiddemann W, Maschmeyer G, Volkers B, et al. Follow-up of the first two successive German multicentre trials for adult ALL (01/81 and 02/84). German Adult ALL Study Group. Leukemia. 1993 Aug;7 Suppl 2:S130-4. No abstract available. PMID 8361217
- [Background] Fiere D, Lepage E, Sebban C, Boucheix C, Gisselbrecht C, Vernant JP, Varet B, Broustet A, Cahn JY, Rigal-Huguet F, et al. Adult acute lymphoblastic leukemia: a multicentric randomized trial testing bone marrow transplantation as postremission therapy. The French Group on Therapy for Adult Acute Lymphoblastic Leukemia. J Clin Oncol. 1993 Oct;11(10):1990-2001. doi: 10.1200/JCO.1993.11.10.1990. PMID 8410124
- [Background] Durrant IJ, Richards SM. Results of Medical Research Council trial UKALL IX in acute lymphoblastic leukaemia in adults: report from the Medical Research Council Working Party on Adult Leukaemia. Br J Haematol. 1993 Sep;85(1):84-92. doi: 10.1111/j.1365-2141.1993.tb08649.x. PMID 8251413
- [Background] Dekker AW, van't Veer MB, Haak HL, van der Lelie J, Ossenkoppele G, Schouten HC, et al. Conventional induction remission followed by intensive consolidation without maintenance therapy in adult acute lymphoblastic leukemia. Results from a phase II in 130 patients. Blood 1994; 84 (suppl 1) 144a.
- [Background] Kantarjian HM, O'Brien S, Smith T, Estey EH, Beran M, Preti A, Pierce S, Keating MJ. Acute lymphocytic leukaemia in the elderly: characteristics and outcome with the vincristine-adriamycin-dexamethasone (VAD) regimen. Br J Haematol. 1994 Sep;88(1):94-100. doi: 10.1111/j.1365-2141.1994.tb04982.x. PMID 7803263
- [Background] Preti HA, Huh YO, O'Brien SM, Andreeff M, Pierce ST, Keating M, Kantarjian HM. Myeloid markers in adult acute lymphocytic leukemia. Correlations with patient and disease characteristics and with prognosis. Cancer. 1995 Nov 1;76(9):1564-70. doi: 10.1002/1097-0142(19951101)76:93.0.co;2-1. PMID 8635059
- [Background] Larson RA, Dodge RK, Burns CP, Lee EJ, Stone RM, Schulman P, Duggan D, Davey FR, Sobol RE, Frankel SR, et al. A five-drug remission induction regimen with intensive consolidation for adults with acute lymphoblastic leukemia: cancer and leukemia group B study 8811. Blood. 1995 Apr 15;85(8):2025-37. PMID 7718875
- [Background] Mandelli F, Annino L, Rotoli B. The GIMEMA ALL 0183 trial: analysis of 10-year follow-up. GIMEMA Cooperative Group, Italy. Br J Haematol. 1996 Mar;92(3):665-72. doi: 10.1046/j.1365-2141.1996.00394.x. PMID 8616033
- [Background] Chessells JM, Bailey C, Richards SM. Intensification of treatment and survival in all children with lymphoblastic leukaemia: results of UK Medical Research Council trial UKALL X. Medical Research Council Working Party on Childhood Leukaemia. Lancet. 1995 Jan 21;345(8943):143-8. doi: 10.1016/s0140-6736(95)90164-7. PMID 7823668
- [Background] JJ Ortega. Tratamiento de las leucemias agudas linfoblásticas del niño. Problemas actuales. En: J Maldonado, ed. Libro de Ponencias. XXXVIII Reunión Nacional de la Asociación Española de Hematología y Hemoterapia. 1996; 175-182.
- [Background] JM Ribera. Quimioterapia de la leucemia aguda linfoblástica del adulto. En: Libro de Ponencias. En: J Maldonado, ed. Libro de Ponencias. XXXVIII Reunión Nacional de la Asociación Española de Hematología y Hemoterapia. 1996; 183-190
- [Background] Schorin MA, Blattner S, Gelber RD, Tarbell NJ, Donnelly M, Dalton V, Cohen HJ, Sallan SE. Treatment of childhood acute lymphoblastic leukemia: results of Dana-Farber Cancer Institute/Children's Hospital Acute Lymphoblastic Leukemia Consortium Protocol 85-01. J Clin Oncol. 1994 Apr;12(4):740-7. doi: 10.1200/JCO.1994.12.4.740. PMID 8151317
- [Background] Rivera GK, Raimondi SC, Hancock ML, Behm FG, Pui CH, Abromowitch M, Mirro J Jr, Ochs JS, Look AT, Williams DL, et al. Improved outcome in childhood acute lymphoblastic leukaemia with reinforced early treatment and rotational combination chemotherapy. Lancet. 1991 Jan 12;337(8733):61-6. doi: 10.1016/0140-6736(91)90733-6. PMID 1670723
- [Background] Reiter A, Schrappe M, Ludwig WD, Hiddemann W, Sauter S, Henze G, Zimmermann M, Lampert F, Havers W, Niethammer D, et al. Chemotherapy in 998 unselected childhood acute lymphoblastic leukemia patients. Results and conclusions of the multicenter trial ALL-BFM 86. Blood. 1994 Nov 1;84(9):3122-33. PMID 7949185
- [Background] Hoelzer D. Critical evaluation of chemotherapy and transplantation of hematopoietic precursor cells in adult ALL. En: J Maldonado, ed. Libro de Ponencias. XXXVIII Reunión Nacional de la Asociación Española de Hematología y Hemoterapia. 1996; 191-193.
- [Background] JM Ribera, JJ Ortega, A Oriol, M Fontanillas, J Maldonado, R Parody, C Rivas, JM Hernández-Rivas, MJ Terol, P Bastida, ME González-Valentín, E Feliu, J García-Conde, J Díaz-Mediavilla, JF san Miguel. Treatment of high-risk acute lymphoblastic leukemia (HRALL). Preliminary results of the protocol PETHEMA ALL-93. Acute Leukemias VII. Experimental Approaches and Novel Therapies. Ann Hematol 1997; 74 (suppl1): A41.
- [Background] Chessells JM, Bailey C, Wheeler K, Richards SM. Bone marrow transplantation for high-risk childhood lymphoblastic leukaemia in first remission: experience in MRC UKALL X. Lancet. 1992 Sep 5;340(8819):565-8. doi: 10.1016/0140-6736(92)92103-m. PMID 1355153
- [Background] von Bueltzingsloewen A, Esperou-Bourdeau H, Souillet G, Demeocq F, Mechinaud-Lacroix F, Michel G, Sadoun A, Bernaudin F, Cornu G, Donadieu J, et al. Allogeneic bone marrow transplantation following a busulfan-based conditioning regimen in young children with acute lymphoblastic leukemia: a Cooperative Study of the Societe Francaise de Greffe de Moelle. Bone Marrow Transplant. 1995 Oct;16(4):521-7. PMID 8528167
- [Background] Saarinen UM, Mellander L, Nysom K, Ringden O, Schroeder H, Glomstein A, Gustafsson G. Allogeneic bone marrow transplantation in first remission for children with very high-risk acute lymphoblastic leukemia: a retrospective case-control study in the Nordic countries. Nordic Society for Pediatric Hematology and Oncology (NOPHO). Bone Marrow Transplant. 1996 Mar;17(3):357-63. PMID 8704687
- [Background] Ortega JJ, Olivé T, Diaz de Heredia C, et al. Allogeneic and autologous bone amrrow transplant in acute lymphoblastic leukaemia. Bone Marrow Transplant 1996; 17 (supl 1): 76
- [Background] Attal M, Blaise D, Marit G, Payen C, Michallet M, Vernant JP, Sauvage C, Troussard X, Nedellec G, Pico J, et al. Consolidation treatment of adult acute lymphoblastic leukemia: a prospective, randomized trial comparing allogeneic versus autologous bone marrow transplantation and testing the impact of recombinant interleukin-2 after autologous bone marrow transplantation. BGMT Group. Blood. 1995 Aug 15;86(4):1619-28. PMID 7632972
- [Background] Barrett AJ. Bone marrow transplantation for acute lymphoblastic leukaemia. Baillieres Clin Haematol. 1994 Jun;7(2):377-401. doi: 10.1016/s0950-3536(05)80209-4. PMID 7803908
- [Background] De Witte T, Awwad B, Boezeman J, Schattenberg A, Muus P, Raemaekers J, Preijers F, Strijckmans P, Haanen C. Role of allogenic bone marrow transplantation in adolescent or adult patients with acute lymphoblastic leukaemia or lymphoblastic lymphoma in first remission. Bone Marrow Transplant. 1994 Nov;14(5):767-74. PMID 7889010
- [Background] Schiller G, Feig SA, Territo M, Wolin M, Lill M, Belin T, Hunt L, Nimer S, Champlin R, Gajewski J. Treatment of advanced acute leukaemia with allogeneic bone marrow transplantation from unrelated donors. Br J Haematol. 1994 Sep;88(1):72-8. doi: 10.1111/j.1365-2141.1994.tb04979.x. PMID 7803259
- [Background] Mehta J, Powles R, Horton C, Milan S, Treleaven J, Tait D, Catovsky D. Bone marrow transplantation for primary refractory acute leukaemia. Bone Marrow Transplant. 1994 Sep;14(3):415-8. PMID 7994265
- [Background] Powles R, Mehta J, Singhal S, Horton C, Tait D, Milan S, Pollard C, Lumley H, Matthey F, Shirley J, et al. Autologous bone marrow or peripheral blood stem cell transplantation followed by maintenance chemotherapy for adult acute lymphoblastic leukemia in first remission: 50 cases from a single center. Bone Marrow Transplant. 1995 Aug;16(2):241-7. PMID 7581142
- [Background] Dicke KA, Hoelzer DF, Gorin NC, Lowenberg B, Gale RP. The role of bone marrow transplantation in adult acute lymphocytic leukemia. Ann Oncol. 1993;4 Suppl 1:81-90. doi: 10.1093/annonc/4.suppl_1.s81. No abstract available. PMID 8338797
- See also: Spanish association of Haematology — http://www.aehh.org